CLINICAL TRIAL: NCT06623851
Title: Effectiveness of Digital Versus Conventional Impression on Discomfort and Dental Anxiety in Preschool Children (A Randomized Controlled Clinical Trial)
Brief Title: Digital Versus Conventional Impression on Discomfort and Dental Anxiety Among Preschoolers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0863-2/2024
Record Dates: First submitted 2024-07-25; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Dental Anxiety
Keywords: Dental impression; Digital impression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital dental Impression (Experimental)
  Interventions: Other: Intraoral scanner
- Conventional dental impression (Active Comparator)
  Interventions: Other: Alginate impression

INTERVENTIONS:
Other: Intraoral scanner — * The digital impressions will be made with the intraoral scanner following the procedure reported by the manufacturer.
  * The intraoral scanning process is divided into the lower jaw scan, upper jaw scan, and bite scan stages
  Arms: Digital dental Impression
Other: Alginate impression — Conventional impressions of both arches will be made according to the manufacturer's instructions, using steel impression trays and alginate
  Arms: Conventional dental impression

SUMMARY:
Background: Taking alginate impressions for preschoolers is challenging and might be disturbing for them. Therefore, intraoral scanners are suggested as a better alternative to the conventional alginate impression.

Objectives: The present study aims to evaluate and compare the level of patients' discomfort, dental anxiety, gag reflex, behavior and time required for taking alginate impressions with that of intraoral scanning.

Materials and methods: The study will be a randomized, controlled clinical trial, parallel design. A total of 666 pediatric dental patients aged from 4-6 years will be selected from the outpatient clinic of the of Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Alexandria University. Participants will be allocated into 2 groups. Children in the first group will receive digital impressions by an intraoral scanner, while those of the second group will receive conventional alginate impressions. Patients' discomfort will be evaluated by a modified VAS index supported with emojis. Dental anxiety will be evaluated using Facial Image Scale (FIS). Gag reflex will be assessed by Gag Severity Index (GSI). Child's behavior towards the impression technique in the 2 groups will be evaluated using Venham's Behavior rating scale. Time taken to complete the procedures will be recorded using a digital stopwatch.

ELIGIBILITY:
Inclusion Criteria:

* Children with scores of 3 or 4 during preoperative assessments according to the Frankl Behavioral Rating Scale.
* No previous dental experience.
* Patient's parents signed an informed consent before participating in the trial.

Exclusion Criteria:

* Any physical or mental disability, or psychological problems.
* Children with temporomandibular joint or periodontal discomfort

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2024-06-23 (Actual); Primary Completion 2024-09-29 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in child discomfort | intraoperative
  Children's discomfort will be evaluated using a 100-mm modified VAS index supported with facial emojis.
Change in dental anxiety | intraoperative
  Dental anxiety will be recorded using the Facial Image Scale (FIS) Children will be asked to indicate which of the faces they feel most like at that moment, it is a 'state' measure of anxiety that provides an immediate reflection of how the child is feeling.

SECONDARY OUTCOMES:
Gag reflex | post procedure
  After taking the impressions, child's gag reflex will be assessed. Gag sensitivity is ranked on a scale from 1 (least severe) to 5 (most severe) using the Gagging Severity Index (GSI)
Assessment of level of child cooperation | intraoperative
  Venham's Behavior rating scale classifies the child's behavior into 6 categories with scores ranging from 0 to 5. A score of 0 means total cooperation and a score of 5 refers to complete absence of compliance and cooperation and the requirement of physical restraint
procedure time | intraoperative
  Time taken from scanning and taking impression for the lower and upper jaws to the final bite registeration. Time will be recorded in minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt